CLINICAL TRIAL: NCT04914819
Title: Postpartum Weight Loss for Women at Elevated Cardiovascular Risk (EmPOWER-Mom Study)
Brief Title: Postpartum Weight Loss for Women at Elevated Cardiovascular Risk
Acronym: EMPOWER-Mom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jennifer Lewey, MD, MPH, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 844694; 5K23HL153667-03 (NIH)
Record Dates: First submitted 2021-05-20; First posted 2021-06-07 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Weight Loss; Postpartum Weight Retention; Hypertension in Pregnancy; Diabetes Mellitus in Pregnancy; Preeclampsia; Recruitment
Keywords: weight loss; postpartum period; hypertension in pregnancy; cardiovascular risk reduction; diabetes prevention program
MeSH Terms: conditions — Weight Loss; Gestational Weight Gain; Hypertension, Pregnancy-Induced; Diabetes, Gestational; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Behavioral Weight Loss (Active Comparator): Participants will attend a virtual introduction to weight loss session and be enrolled in a 16-week online behavioral weight loss program. Participants will complete a virtual weigh-in at the start and end of the study.
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual weigh-in
- Usual Care (Active Comparator): Participants will complete a virtual weigh-in at the start and end of the study. No additional intervention will be provided.
  Interventions: Behavioral: Virtual weigh-in

INTERVENTIONS:
Behavioral: Online Behavioral Weight Loss Program — Participants will be enrolled in a 16-week online behavioral weight loss program based on the Diabetes Prevention Program (DPP). The program involves weekly brief videos, a self-monitoring platform, automated feedback, and access to a health coach.
  Arms: Online Behavioral Weight Loss
Behavioral: Virtual weigh-in — Participants will be sent a digital scale and will be asked to complete a virtual weigh-in at home at the start of the study and again after 16 weeks.

SUMMARY:
The aim of this study is to test the feasibility and effectiveness of a 16-week online behavioral weight loss program compared to usual care to promote weight loss in the postpartum period among women with cardiovascular risk factors. The investigators will also be testing different behavioral strategies to recruit postpartum women to the study, including 2 email recruitment strategies and 2 mailer recruitment strategies, informed by behavioral design.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Delivered a baby at HUP or PAH within 3-12 months prior to study start;
3. BMI ≥ 27 kg/m2
4. Diagnosis of one of the following medical conditions: chronic hypertension, gestational hypertension, preeclampsia, eclampsia, gestational diabetes, or diabetes mellitus (type 1 or 2) based on diagnosis codes in the EMR
5. Has online access through smartphone or computer and has email address
6. Ability to read and provide informed consent to participate in the study

Exclusion Criteria:

1. Delivered prior to 32 weeks gestation in the EMR
2. Documentation of fetal demise or neonatal demise in the EMR
3. Currently pregnant or planning to get pregnant within the next 5 months
4. Does not speak English
5. Answers yes to any of the following questions:

   * Are you currently participating in any other weight loss or physical activity studies?
   * Do you have any medical conditions or other reasons why you could not participate in a 16-week weight loss or physical activity program?
6. Participants will be excluded after completing the run-in period if they do not complete the daily food log or their baseline BMI is < 27 kg/m2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,047 participants were invited to participate in the study. Potentially eligible participants were recruited from the electronic health record and were sent an email invitation (n=1,000). Potentially eligible participants who did not respond to email recruitment and those who did not have an email address also received a mailer recruitment letter (n=849).
Pre-assignment Details: 190 individuals signed up for an info session.
  Of the 190, 115 attended the info session. Excluded: 75 individuals did not attend info session.
  Of the 115, 89 provided consent and enrolled in run-in period. Excluded: 26 individuals who did not provide consent.
  Of the 89 enrolled, 60 completed run-in period and were randomized to one of two arms.
  Note: 27 people signed up for an info session after receiving a recruitment mailer but were excluded due to recruitment goals being met.
Period: Overall Study
Arm/Group | Online Behavioral Weight Loss | Usual Care
Started | 40 | 20
Completed | 26 | 18
Not Completed | 14 | 2
Not completed — Pregnancy | 3 | 1
Not completed — Discontinued study | 4 | 1
Not completed — Lost to Follow-up | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Behavioral Weight Loss | Usual Care | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0
  Age: Between 18 and 65 years | 40 | 20 | 60
  Age: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (5.7) | 32 (4.2) | 33.1 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 20 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 37 | 18 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 10 | 29
  White | 19 | 8 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60
Chronic hypertension [Count of Participants; unit: Participants] | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight in Pounds From Baseline to 16-week Follow-up
Description: Mean change in weight in pounds from baseline to 16-week follow-up between study arms.
Time Frame: Baseline and 16 weeks
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Online Behavioral Weight Loss | Usual Care
Number analyzed (Participants) | 40 | 20
pounds | -8.6 [-12.1 to -5.3] | -3.3 [-7.3 to -0.9]
Statistical Analysis 1: Comparison: Online Behavioral Weight Loss vs Usual Care; Change in weight among participants who completed final assessment; Test type: Superiority; p = 0.048, Mixed Models Analysis; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [0.04 to 10.8]

2. Primary Outcome: Enrollment Rate Between Email Recruitment Strategies
Description: We will compare enrollment rates between two behaviorally-framed email strategies
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Email 1: Reserved a Spot: Individuals were recruited via email using a standard script that ended with: "We saved a spot just for you at our on-line information session. Click below to learn more. Don't give away my spot!"
- Email 2: Commit to Health: Individuals were recruited via email using a standard script that ended with: "Are you ready to commit to your own health? Space is limited, so sign-up before all the spots are gone. I am ready to commit."
Arm/Group | Email 1: Reserved a Spot | Email 2: Commit to Health
Number analyzed (Participants) | 497 | 503
Participants | 88 | 102
Statistical Analysis 1: Comparison: Email 1: Reserved a Spot vs Email 2: Commit to Health; Test type: Superiority; p = 0.3, Chi-squared

3. Primary Outcome: Sign-up Rate Between Mailer Recruitment Strategies
Description: We will compare enrollment rates between the group receiving a mailer versus mailer plus baby gift
Time Frame: 8 weeks
Population: A total of 849 patients were randomized to one of two mailer strategies. Participants were eligible for randomization if they met eligibility criteria in the EHR and did not respond to the email invitation (either signed up for information session or declined invitation). They were also eligible for randomization if they had a mailing address but did not have an email address on file.
Measure: Count of Participants; unit: Participants
Groups:
- Mailer Alone: Individuals who did not respond to the initial recruitment email were sent a mailer with more study information. We also included participants who did not have a documented email in the EHR.
- Mailer + Gift: Individuals who did not respond to the initial recruitment email were sent a mailer with more study information and a gift. We also included participants who did not have a documented email in the EHR.
Arm/Group | Mailer Alone | Mailer + Gift
Number analyzed (Participants) | 424 | 425
Participants | 11 | 16
Statistical Analysis 1: Comparison: Mailer Alone vs Mailer + Gift; Test type: Superiority; p = 0.331, Chi-squared

4. Primary Outcome: Number of Participants Losing 5 Percent or More of Weight From Baseline to 16-week Follow-up
Description: Proportion of participants who lost 5 percent or more of their weight from baseline to 16-week follow-up between study groups.
Time Frame: Baseline and 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Online Behavioral Weight Loss | Usual Care
Number analyzed (Participants) | 40 | 20
Participants | 9 | 3
Statistical Analysis 1: Comparison: Online Behavioral Weight Loss vs Usual Care; Test type: Superiority; p = 0.734, Fisher Exact

5. Secondary Outcome: Study Completion Rate Between 2 Arms
Description: Proportion of participants that completed all follow-up procedures between both study arms.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Online Behavioral Weight Loss | Usual Care
Number analyzed (Participants) | 40 | 20
Participants
  Completed follow-up | 26 | 18
  Discontinued intervention | 4 | 1
  Pregnant | 3 | 1
  Lost to follow-up | 7 | 0

6. Secondary Outcome: Intervention Arm: Number of Weeks With One or More Logins
Description: Engagement with BWL platform measured by mean number of weeks with one or more logins
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Online Behavioral Weight Loss
Number analyzed (Participants) | 40
weeks | 8.6 (5.3)

7. Secondary Outcome: Intervention Arm: Number of Weeks With Daily Data Reporting for at Least 5 of 7 Days
Description: Mean number of weeks that calories, physical activity minutes, and body weight were reported at least 5 of 7 days
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Online Behavioral Weight Loss
Number analyzed (Participants) | 40
weeks | 5.2 (4.8)

ADVERSE EVENTS:
Time Frame: 1-week behavioral run-in plus 16 weeks intervention
Description: Standard definitions were used
Groups:
- Run-In Phase: Participants who provide consent will be asked to complete a 7 day "run-in phase" where they are asked to track their meals daily in the online meal tracker app or on paper. After completing this period, participants are eligible to be randomized.
Arm/Group | Online Behavioral Weight Loss | Usual Care | Run-In Phase
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20 | 0/89
Other Adverse Events (participants affected / at risk) | 0/40 | 0/20 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT04914819/Prot_SAP_000.pdf